CLINICAL TRIAL: NCT01117194
Title: Rehabilitation Robot for Upper Limbs, Component Project 5: Effect on Shoulder Training Using Rehabilitation Robot for Stroke Patients
Brief Title: Effect on Shoulder Training Using Rehabilitation Robot for Stroke Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 200804031D
Record Dates: First submitted 2010-01-18; First posted 2010-05-05 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- shoulder training, rehabilitation robot (Experimental)
  Interventions: Device: Rehabilitation Robot for Upper Limb Dysfunction (NTUH Model One)
- control group (No Intervention)

INTERVENTIONS:
Device: Rehabilitation Robot for Upper Limb Dysfunction (NTUH Model One) — Use an intelligent robot to assist upper limb rehabilitation.
  Other Names: self-developed robotic arm
  Arms: shoulder training, rehabilitation robot

SUMMARY:
The purpose is to study the effect of rehabilitation robot on shoulder training for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* stroke (1-3 months)
* Brunnstrom Stage II-III
* single, unilateral

Exclusion Criteria:

* aphasic
* shoulder impairment
* severe osteoporosis

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Barthel index, | 1 year
Modified Asworth Scale | 1 year
STREAM and PASS scales | 1 year

SECONDARY OUTCOMES:
shoulder range of motion, VAS | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Shiang Chen, MD, PhD, Principal Investigator — Dpt. Physical Medicine and Rehabilitation, NTUH Taipei, Taiwan
Locations (1):
- Dpt. Physical Medicine and Rehabilitation, NTUH, Taipei, Taiwan